CLINICAL TRIAL: NCT02813733
Title: Influence of Factors Specific to Patient, Procedure or Surgeon on Thyroid Surgery Outcomes
Brief Title: Determinants of Thyroid Surgery Outcomes
Acronym: CATHY
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50528
Record Dates: First submitted 2016-06-22; First posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Thyroid Disease
Keywords: thyroid surgery; surgical outcomes; patient safety; healthcare quality; surgeons performance
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thyroid surgery: All patients who underwent a thyroid procedure in 5 high volume referral centers in France were eligible for inclusion.
  Interventions: Procedure: Thyroid surgery

INTERVENTIONS:
Procedure: Thyroid surgery — Thyroidectomies performed by all surgeons in 5 academic hospitals in France.

SUMMARY:
In a large prospective cross-sectional study, the investigators aimed to identify the determinants of thyroid surgery outcomes and quantify the relative influence of preoperative and intraoperative factors. For this purpose, the investigators considered the interplay of several characteristics specific to surgeons, patients, and surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

- All patients who underwent a thyroid procedure between April 2008 and July 2008.

Exclusion Criteria:

- Participation refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent a thyroid procedure during study period in 5 high volume referral centers in France were eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Recurrent laryngeal nerve palsy | During inpatient stay and at 6 months following surgery
  Systematic postoperative screening by laryngoscopy

SECONDARY OUTCOMES:
Secondary hypoparathyroidism | During inpatient stay and at 6 months following surgery
  Systematic postoperative screening based on hypocalcaemia < 2 mmoL/l or vitaminocalcic substitution

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Lifante, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon - Centre Hospitalier Lyon Sud, 165 Chemin du Grand Revoyet, Pierre-Bénite, France